CLINICAL TRIAL: NCT03660592
Title: Contribution LUS and Reproducibility of Lung Ultrasound in the Diagnosis of Acute Heart Failure in the Emergency Department (ED)
Brief Title: Contribution and Reproducibility of Lung Ultrasound in the Diagnosis of Acute Heart Failure in the ED
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Pr Nouira Semir, University of Monastir
Other Study IDs: LUS/HF
Record Dates: First submitted 2018-07-06; First posted 2018-09-06 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Dyspnea; Cardiac
Keywords: Lung ultrasound; heart failure; diagnosis
MeSH Terms: conditions — Dyspnea; Heart Failure; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- operator 1: ED resident experimented in pulmonary ultrasonography and blinded to the final diagnosis
- operator 2: a different ED resident experimented in pulmonary ultrasonography and blinded to the final diagnosis

SUMMARY:
Discrimination between cardiac and non-cardiac causes of dyspnea can be challenging, causing excessive delay before adequate therapy. In clinical practice lung ultrasound (LUS) is becoming an easy and reliable noninvasive tool for the evaluation of dyspnea and can shorten the time to diagnosis .However the reproductibility of this test was not extensively studied.

DETAILED DESCRIPTION:
Dyspnea is one of the most distressing situations for the patient . Emergency cases do not always present in conditions that are ideal for immediate diagnosis, which sometimes compromises outcome. Physical examination, laboratory findings and radiography are imperfect, resulting in a need for sophisticated test results that delay management.

Lung ultrasonography is becoming a standard tool in critical cases in the ED.

the investigators aim to perform ultrasonography on consecutive patients admitted to the ICU with dyspnea, comparing lung ultrasonography results on initial presentation with the final diagnosis by the ICU team.

Three items were assessed: artifacts (horizontal A lines or vertical B lines indicating interstitial syndrome), lung sliding, and alveolar consolidation and/or pleural effusion, these items were grouped to assess ultrasound profiles.

This study assesses the potential of lung ultrasonography to diagnose heart failure.The second aim of this study was to evaluate the inter-observer reproducibility of LUS performed by ED residents in the evaluation of cardiac causes of acute dyspnea.

Patients presenting to the ED with acute dyspnea will be prospectively enrolled in this study. In each patient, LUS was performed by two ED residents blinded to clinical diagnoses.

AHF was determined on the base of clinical exam, chest x-ray , brain natriuretic peptide (BNP) and echocardiographic findings.

A patient lung comet score (LCS) was obtained by summing the number of comets in each of the scanned spaces.

Then the probability of AHF was defined as :

low probability (LCS<15) intermediate probability (15 <LCS<30), and high probability (LCS>30 ).

ELIGIBILITY:
Inclusion Criteria:

* non traumatic dyspnea with the final diagnosis of heart failure

Exclusion Criteria:

* impossibility to give consent to participate in the study
* post traumatic dyspnea
* pregnant women
* need for endotracheal intubation or inotropic drugs
* patients who were deemed too unstable for sonography by the treating team

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients admitted to the ED with acute dyspnea, with the final diagnosis of heart failure
Sampling Method: Non-Probability Sample
Enrollment: 1024 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
the reproductibility of LUS in the diagnosis of heart failure | 0 days
  the reproductibility of the LUS in the diagnosis of heart failure between two different operators (using the Kappa and the agreement index)
the accuracy of LUS in the diagnosis of heart failure the accuracy of LUS in the diagnosis of heart failure measured by sensitivity ,specificity, and area under the roc curve | 0 days
  the accuracy of LUS in the diagnosis of heart failure measured by sensitivity ,specificity, and area under the roc curve

CONTACTS AND LOCATIONS:
Overall Officials: Nouira semir, professor, Principal Investigator — university of ùmonastir

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: official department website — http://www.urgencemonastir.com